CLINICAL TRIAL: NCT05672381
Title: Near-infrared Spectroscopic Tomography (NIRST) and ICG-based Perfusion Imaging to Diagnose and Assess Muscle Viability in High Energy Trauma at Risk for Acute Compartment Syndrome: A Pilot Study
Brief Title: NIRST and ICG-based Perfusion Imaging in Acute Compartment Syndrome
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: Dartmouth College (Other)
Responsible Party: Principal Investigator, Ida Leah Gitajn, Section Chief, Dartmouth-Hitchcock Medical Center
Other Study IDs: STUDY02001595
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2024-09

CONDITIONS: Compartment Syndromes; Compartment Syndrome of Lower Leg; Compartment Syndrome of Forearm
MeSH Terms: conditions — Compartment Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Lower leg Trauma: High-energy lower leg trauma at risk for Acute Compartment Syndrome
  Interventions: Procedure: Lower extremity and/or upper extremity surgery
- Forearm Trauma: High-energy forearm trauma at risk for Acute Compartment Syndrome
  Interventions: Procedure: Lower extremity and/or upper extremity surgery

INTERVENTIONS:
Procedure: Lower extremity and/or upper extremity surgery — Lower extremity and/or upper extremity surgery

SUMMARY:
This is a prospective observational study of patients with suspected Acute Compartment Syndrome. The primary objective of this work is to determine whether intensity changes associated with the NIRST signal, reflecting oxy- and deoxy-hemaglobin and water concentrations or ICG fluorescence signal, reflecting tissue perfusion, can be associated with development of Acute Compartment Syndrome and identification of at-risk soft tissue and muscle.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Clinical suspicion of acute compartment syndrome based on orthopaedic provider assessment. Clinical suspicion would be based upon the presence of one or more of these findings:

  * Pain out of proportion to visible findings
  * Escalating doses of pain medication
  * Pain with passive stretch of toes and/or fingers
  * Pallor, paresthesias, pulselessness
  * Tense soft tissues
  * High energy tibia or forearm fracture
* Provision of informed consent

Exclusion Criteria:

* History of allergy to ICG and/or iodine
* Pregnant women or nursing mothers
* Any patient with an open wound for whom NIRST device cannot be applied >4cm from the open wound will be excluded from NIRST imaging.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects receiving care at DHMC (Lebanon) with high energy lower leg or forearm trauma at risk for Acute Compartment Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2025-09-16 (Actual); Study Completion 2025-09-16 (Actual)

PRIMARY OUTCOMES:
Association of NIRST or ICG measurements with development of ACS | 36 months
  The primary objective of this work is to determine whether total hemoglobin, oxygen saturation and water content imaged by NIRST or ICG fluorescence signal, reflecting tissue perfusion, can be associated with development of Acute Compartment Syndrome and identification of at-risk soft tissue and muscle.

CONTACTS AND LOCATIONS:
Overall Officials: Ida L Gitajn, MD, MS, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No